CLINICAL TRIAL: NCT00761631
Title: A Phase 3, Open Label Trial Evaluating the Safety,Tolerability and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine in Healthy Children Aged 15 Months to 17 Years in the United States
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine (13vPnC) in Healthy Children Aged 15 Months to 17 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3011
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): Open label
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13 valent pneumococcal conjugate vaccine — Intramuscular injection of 0.5mL at visit 1 and visit 2 for group 1 and and visit 1 for groups 2, 3, and 4.

SUMMARY:
This open-label, multicenter study is designed to evaluate the safety, tolerability and immunogenicity of 13-valent pneumococcal conjugate vaccine in healthy children aged more than 15 months up to less than 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >15months to <18years in good health, available for entire study period and reachable by phone, parents/legal guardian able and willing to complete all study procedures, written documentation from health professional showing prior vaccination with Prevnar (except for group 4).

Group 4 only:

* Negative urine pregnancy test for female subjects who are menstruating.

Exclusion Criteria:

* Previous reaction or contra-indication to pneumococcal vaccine or vaccine related component , bleeding diathesis, received blood transfusion or blood related products, immune deficiency,congenital malformation.

Group 4 only:

* Previous vaccination with Prevnar or any other pneumococcal vaccine.
* Pregnant or breastfeeding adolescent females.

Ages: 15 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (31):
  - Pfizer Investigational Site, Benton, Arkansas
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, DeKalb, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Whitehouse Station, New Jersey
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Clarksville, Tennessee
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, South Jordan, Utah
  - Pfizer Investigational Site, Vienna, Virginia
  - Pfizer Investigational Site, Vancouver, Washington
  - Pfizer Investigational Site, Monroe, Wisconsin

REFERENCES:
- [Derived] Frenck R Jr, Thompson A, Senders S, Harris-Ford L, Sperling M, Patterson S, Devlin C, Jansen KU, Gruber WC, Emini EA, Scott DA, Gurtman A. 13-Valent pneumococcal conjugate vaccine in older children and adolescents either previously immunized with or naive to 7-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2014 Feb;33(2):183-9. doi: 10.1097/INF.0000000000000056. PMID 24136369
- [Derived] Frenck R Jr, Thompson A, Yeh SH, London A, Sidhu MS, Patterson S, Gruber WC, Emini EA, Scott DA, Gurtman A; 3011 Study Group. Immunogenicity and safety of 13-valent pneumococcal conjugate vaccine in children previously immunized with 7-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2011 Dec;30(12):1086-91. doi: 10.1097/INF.0b013e3182372c6a. PMID 21983216
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3011&StudyName=Study%20Evaluating%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20in%20Healthy%20Children%20Aged%2015%20months%20to%2017%20Years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified by age group. Group 1 included participants aged greater than (>) 15 months to less than (<) 2 years. Group 2 included participants aged greater than or equal to (>=) 2 to <5 years. Group 3 included participants aged >=5 to <10 years. Group 4 included participants aged >=10 to <18 years.
Groups:
- 13vPnC Group 1 (Cohort 1): 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly at baseline and anytime from Day 56 to Day 70 for a total of 2 doses. Participants must have previously received at least 3 doses of 7-valent pneumococcal conjugate vaccine (7vPnC). Includes participants enrolled prior to protocol amendment to increase sample size (Cohort 1).
- 13vPnC Group 2 (Cohort 1): 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to protocol amendment to increase sample size (Cohort 1).
- 13vPnC Group 1 (Cohort 2): 13vPnC (0.5mL dose) administered intramuscularly at baseline and anytime from Day 56 to Day 70 for a total of 2 doses. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled after protocol amendment to increase sample size (Cohort 2).
- 13vPnC Group 2 (Cohort 2): 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled after protocol amendment to increase sample size (Cohort 2).
- 13vPnC Group 3: 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 1 dose of 7vPnC.
- 13vPnC Group 4: 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must not have received 7vPnC or any other pneumococcal vaccine.
Period: Overall Study
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 2 (Cohort 1) | 13vPnC Group 1 (Cohort 2) | 13vPnC Group 2 (Cohort 2) | 13vPnC Group 3 | 13vPnC Group 4
Started | 126 | 181 | 176 | 119 | 299 | 299
Vaccinated Dose 1 | 124 | 179 | 175 | 118 | 294 | 298
Vaccinated Dose 2 | 112 | 0 | 165 | 0 | 0 | 0
Completed | 111 | 174 | 160 | 116 | 277 | 294
Not Completed | 15 | 7 | 16 | 3 | 22 | 5
Not completed — Parent/legal guardian request | 8 | 3 | 8 | 0 | 5 | 0
Not completed — Lost to Follow-up | 2 | 4 | 7 | 1 | 6 | 1
Not completed — Protocol Violation | 2 | 0 | 0 | 1 | 5 | 1
Not completed — Randomized, not treated | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to return | 1 | 0 | 1 | 1 | 5 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC Group 1 (Cohort 1 and 2): 13vPnC (0.5mL dose) administered intramuscularly at baseline and anytime from Day 56 to Day 70 for a total of 2 doses. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to and after protocol amendment to increase sample size (Cohort 1 and Cohort 2, combined)
- 13vPnC Group 2 (Cohort 1 and 2): 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to and after protocol amendment to increase sample size (Cohort 1 and Cohort 2, combined)
- Total: Total of all reporting groups
Arm/Group | 13vPnC Group 1 (Cohort 1 and 2) | 13vPnC Group 2 (Cohort 1 and 2) | 13vPnC Group 3 | 13vPnC Group 4 | Total
Number analyzed (Participants) | 302 | 300 | 299 | 299 | 1200
Age, Customized [Number; unit: Participants]
  >15 months to <2 years | 302 | 0 | 0 | 0 | 302
  >=2 years to <5 years | 0 | 300 | 0 | 0 | 300
  >=5 years to <10 years | 0 | 0 | 299 | 0 | 299
  >10 years to <18 years | 0 | 0 | 0 | 299 | 299
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 139 | 155 | 136 | 578
  Male | 154 | 161 | 144 | 163 | 622

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Predefined Serotype-specific Immunoglobulin G (IgG) Antibody Concentration Greater Than or Equal to (≥) 0.35 Micrograms Per Milliliter (Mcg/mL) Measured 1 Month After Vaccination in Group 1 and 2
Description: Percentage of participants achieving world health organization (WHO) predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. Exact 2-sided CI based on observed proportion of participants.
Time Frame: 28 to 42 days after dose 2 for Group 1 and 28 to 42 days after dose 1 for Group 2
Population: Evaluable Immunogenicity Population (EIP): all participants who met all inclusion criteria, received all assigned doses of study vaccine, had at least 1 valid and determinate assay result from blood draw within 27-56 days after last scheduled vaccination for proposed analysis and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 13vPnC Group 1 (Cohort 1): 13vPnC (0.5mL dose) administered intramuscularly at baseline and anytime from Day 56 to Day 70 for a total of 2 doses. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to protocol amendment to increase sample size (Cohort 1).
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 2 (Cohort 1)
Number analyzed (Participants) | 109 | 175
Percentage of participants
  Common serotypes - serotype 4 | 98.2 [93.5 to 99.8] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 6B | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 9V | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 14 | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 18C | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 19F | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Common serotypes - serotype 23F | 99.1 [95.0 to 100.0] | 100.0 [97.9 to 100.0]
  Additional serotypes - serotype 1 | 100.0 [96.7 to 100.0] | 98.9 [95.9 to 99.9]
  Additional serotypes - serotype 3 | 94.5 [88.4 to 98.0] | 92.0 [86.9 to 95.5]
  Additional serotypes - serotype 5 | 100.0 [96.7 to 100.0] | 98.9 [95.9 to 99.9]
  Additional serotypes - serotype 6A | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Additional serotypes - serotype 7F | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]
  Additional serotypes - serotype 19A | 100.0 [96.7 to 100.0] | 100.0 [97.9 to 100.0]

2. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Measured 1 Month After Vaccination in Group 3
Description: Antibody GMC for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for after dose 1 blood draw.
Time Frame: 28 to 42 days after dose 1 for Group 3
Population: EIP: participants who met all inclusion criteria, received all assigned doses of study vaccine;had at least 1 valid, determinate assay result from blood draw within 27-56 days after last scheduled vaccination for proposed analysis;no major protocol violations. N (number of participants analyzed)=participants with determinate antibody concentration.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 3
Number analyzed (Participants) | 171
mcg/mL
  Common serotypes - serotype 4 | 8.45 [7.24 to 9.87]
  Common serotypes - serotype 6B | 53.56 [45.48 to 63.07]
  Common serotypes - serotype 9V | 9.51 [8.38 to 10.78]
  Common serotypes - serotype 14 | 29.36 [24.78 to 34.78]
  Common serotypes - serotype 18C | 8.23 [7.13 to 9.51]
  Common serotypes - serotype 19F | 17.58 [14.95 to 20.67]
  Common serotypes - serotype 23F | 11.26 [9.79 to 12.95]
  Additional serotypes - serotype 1 | 3.57 [3.05 to 4.18]
  Additional serotypes - serotype 3 | 2.38 [2.07 to 2.74]
  Additional serotypes - serotype 5 | 5.52 [4.82 to 6.32]
  Additional serotypes - serotype 6A | 21.51 [18.15 to 25.51]
  Additional serotypes - serotype 7F | 6.24 [5.49 to 7.08]
  Additional serotypes - serotype 19A | 17.18 [15.01 to 19.67]

3. Primary Outcome: Comparison of Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Measured 1 Month After 13vPnC Vaccination in Group 3 Relative to Posttoddler Responses in Study 6096A1-3005 (NCT00444457)
Description: Comparison of IgG concentrations 1 month after 13vPnC vaccination in group 3 of study 6096A1-3011 (NCT00761631) to posttoddler responses in 7-valent pneumococcal conjugate vaccine (7vPnC) group for 7 common serotypes and in combined 13vPnC groups for 6 additional serotypes of study 6096A1-3005 (NCT00444457) is not reported here because analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in study and described in Participant Flow and Baseline Characteristics modules.
Time Frame: 28 to 42 days after dose 1
Reporting Status: Not Posted
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL

4. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Vaccination in Group 3 and 4
Description: Serotype-specific OPA GMTs for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were determined in the blood samples of all the participants using a microcolony OPA (mcOPA) assay. GMT (13vPnC) and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for after dose 1 blood draw.
Time Frame: 28 to 42 days after dose 1 for Group 3 and 4
Population: EIP: participants who met all inclusion criteria, received all assigned doses of study vaccine;had at least 1 valid, determinate assay result from blood draw within 27-56 days after last scheduled vaccination for proposed analysis;no major protocol violations. N (number of participants analyzed)=participants with a determinate antibody titer.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 3 | 13vPnC Group 4
Number analyzed (Participants) | 189 | 181
titer
  Common serotypes - serotype 4 | 6912 [6101.2 to 7831.4] | 4629 [4017.2 to 5334.3]
  Common serotypes - serotype 6B | 14224 [12316.4 to 16427.3] | 14996 [13164.1 to 17083.1]
  Common serotypes - serotype 9V | 4485 [4001.1 to 5027.5] | 4733 [4203.3 to 5328.4]
  Common serotypes - serotype 14 | 6894 [6028.3 to 7884.0] | 4759 [4120.4 to 5497.0]
  Common serotypes - serotype 18C | 6263 [5436.4 to 7215.1] | 8815 [7738.2 to 10041.0]
  Common serotypes - serotype 19F | 2280 [1949.4 to 2667.6] | 1559 [1293.3 to 1878.9]
  Common serotypes - serotype 23F | 3808 [3354.7 to 4322.6] | 3245 [2818.8 to 3735.5]
  Additional serotypes - serotype 1 | 319 [271.2 to 376.0] | 187 [160.4 to 218.6]
  Additional serotypes - serotype 3 | 114 [100.4 to 129.4] | 202 [180.9 to 226.3]
  Additional serotypes - serotype 5 | 336 [270.3 to 417.6] | 491 [426.3 to 565.3]
  Additional serotypes - serotype 6A | 9928 [8457.0 to 11654.8] | 7514 [6350.8 to 8890.7]
  Additional serotypes - serotype 7F | 6584 [5829.4 to 7435.5] | 10334 [9099.0 to 11736.8]
  Additional serotypes - serotype 19A | 1276 [1131.7 to 1439.0] | 1180 [1047.5 to 1329.4]
Statistical Analysis 1: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.5, 95% CI 2-sided [1.24 to 1.80]
Statistical Analysis 2: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.9, 95% CI 2-sided [0.78 to 1.15]
Statistical Analysis 3: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.9, 95% CI 2-sided [0.80 to 1.12]
Statistical Analysis 4: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.19 to 1.76]
Statistical Analysis 5: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.7, 95% CI 2-sided [0.59 to 0.86]
Statistical Analysis 6: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.5, 95% CI 2-sided [1.15 to 1.86]
Statistical Analysis 7: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.2, 95% CI 2-sided [0.97 to 1.42]
Statistical Analysis 8: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.7, 95% CI 2-sided [1.36 to 2.13]
Statistical Analysis 9: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.6, 95% CI 2-sided [0.48 to 0.67]
Statistical Analysis 10: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.7, 95% CI 2-sided [0.53 to 0.89]
Statistical Analysis 11: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.3, 95% CI 2-sided [1.05 to 1.67]
Statistical Analysis 12: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.6, 95% CI 2-sided [0.53 to 0.76]
Statistical Analysis 13: Comparison: 13vPnC Group 3 vs 13vPnC Group 4; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC Group 4 - 13vPnC Group 3); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.1, 95% CI 2-sided [0.91 to 1.28]

5. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 7 Days of Dose 1
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm).
Time Frame: From the day of dose 1 (Day 1) to Day 7 after dose 1
Population: Dose 1 Safety Population: all participants who received the first dose of 13vPnC. 'N' (number of participants analyzed )=participants with known values for any local reaction. 'n'=number of participants with known values for specified local reaction for each group respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 2 (Cohort 1) | 13vPnC Group 1 (Cohort 2) | 13vPnC Group 2 (Cohort 2) | 13vPnC Group 3 | 13vPnC Group 4
Number analyzed (Participants) | 110 | 158 | 151 | 102 | 270 | 285
Percentage of participants
  Tenderness Any (n=108,155, 148,102,265,283) | 50.9 | 61.9 | 45.3 | 62.7 | 86.8 | 89.0
  Tenderness Significant (n=92,141,133,92,221,242) | 7.6 | 10.6 | 5.3 | 13.0 | 19.5 | 43.8
  Swelling Any (n=97,144,142,90,226,233) | 25.8 | 22.2 | 17.6 | 20.0 | 37.6 | 36.9
  Swelling Mild (n=94,143,141,89,220,221) | 21.3 | 20.3 | 14.2 | 13.5 | 21.8 | 22.6
  Swelling Moderate (n=94,141,135,89,219,226) | 9.6 | 5.7 | 7.4 | 11.2 | 21.9 | 21.2
  Swelling Severe (n=90,138,131,88,211,214) | 0.0 | 0.0 | 0.0 | 1.1 | 3.3 | 1.9
  Redness Any (n=103,149,143,91,233,232) | 39.8 | 34.9 | 18.9 | 36.3 | 42.9 | 30.2
  Redness Mild (n=99,146,143,90,226,226) | 31.3 | 31.5 | 16.8 | 31.1 | 27.9 | 21.2
  Redness Moderate (n=94,142,135,89,218,221) | 12.8 | 9.9 | 5.9 | 14.6 | 22.0 | 14.0
  Redness Severe (n=90,138,131,88,212,213) | 0.0 | 0.0 | 0.8 | 1.1 | 3.3 | 1.9

6. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 7 Days of Dose 2
Description: as for outcome 5
Time Frame: From the day of dose 2 (Day 1) to Day 7 of dose 2
Population: Dose 2 Safety Population: all participants who received 2 doses of 13vPnC. 'N' (number of participants analyzed )=participants with known values for any local reaction. 'n'=number of participants with known values for specified local reaction for each group respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 1 (Cohort 2)
Number analyzed (Participants) | 90 | 131
Percentage of participants
  Tenderness Any (n=87, 125) | 57.5 | 55.2
  Tenderness Significant (n=68, 101) | 8.8 | 9.9
  Swelling Any (n=73, 105) | 23.3 | 17.1
  Swelling Mild (n=72, 104) | 22.2 | 15.4
  Swelling Moderate (n=69, 102) | 2.9 | 7.8
  Swelling Severe (n=68, 98) | 0.0 | 0.0
  Redness Any (n=76, 110) | 35.5 | 23.6
  Redness Mild (n=74, 108) | 33.8 | 18.5
  Redness Moderate (n=70, 100) | 7.1 | 6.0
  Redness Severe (n=68, 98) | 0.0 | 0.0

7. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Systemic Events Within 7 Days of Dose 1
Description: Systemic events (any fever >=38 degrees [deg] Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary.
Time Frame: From the day of dose 1 (Day 1) to Day 7 of dose 1
Population: Dose 1 Safety Population: all participants who received the first dose of 13vPnC. 'N' (number of participants analyzed )=participants with known values for any systemic events. 'n'=number of participants with known values for specified systemic events for each group respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 2 (Cohort 1) | 13vPnC Group 1 (Cohort 2) | 13vPnC Group 2 (Cohort 2) | 13vPnC Group 3 | 13vPnC Group 4
Number analyzed (Participants) | 112 | 157 | 165 | 107 | 250 | 253
Percentage of participants
  Fever >=38 to <=39 degC(n=92,138,137,90,212,214) | 16.3 | 5.1 | 17.5 | 14.4 | 4.2 | 5.1
  Fever >39 but <=40 degC(n=90,138,130,89,212,212) | 4.4 | 0.7 | 4.6 | 3.4 | 2.4 | 0.5
  Fever >40 degC (n=90,138,130,88,210,212) | 0.0 | 0.7 | 0.0 | 1.1 | 0.5 | 0.5
  Decreased appetite (n=99,149,146,94,227,223) | 42.4 | 24.8 | 39.7 | 34.0 | 22.9 | 22.9
  Irritability (n=108,151,156,102,234,234) | 60.2 | 39.7 | 72.4 | 52.0 | 31.2 | 25.2
  Increased sleep (n=98,145,146,97,226,229) | 32.7 | 15.9 | 37.0 | 23.7 | 21.2 | 26.6
  Decreased sleep (n=97,143,140,91,212,224) | 22.7 | 14.0 | 32.1 | 18.7 | 5.7 | 18.8
  Hives (urticaria) (n=90,139,131,88,213,214) | 1.1 | 0.7 | 1.5 | 4.5 | 1.9 | 1.4

8. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Systemic Events Within 7 Days of Dose 2
Description: Systemic events (any fever >=38 deg C, decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may have been represented in more than 1 category. Percentage of participants = number of participants reporting specified systemic event divided by number of participants reporting yes for at least 1 day or no for all days.
Time Frame: From the day of dose 2 (Day 1) to Day 7 of dose 2
Population: Dose 2 Safety Population: all participants who received 2 doses of 13vPnC. 'N' (number of participants analyzed )=participants with known values for any systemic events. 'n'=number of participants with known values for specified systemic events for each group respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC Group 1 (Cohort 1) | 13vPnC Group 1 (Cohort 2)
Number analyzed (Participants) | 91 | 137
Percentage of participants
  Fever >=38 but <=39 degC (n=70,101) | 14.3 | 11.9
  Fever >39 but <=40 degC (n=68, 100) | 4.4 | 2.0
  Fever >40 degC (n=68, 98) | 0.0 | 1.0
  Decreased appetite (n=77, 113) | 40.3 | 34.5
  Irritability (n=86, 126) | 65.1 | 61.1
  Increased sleep (n=75, 109) | 29.3 | 23.9
  Decreased sleep (n=77, 112) | 28.6 | 26.8
  Hives (urticaria) (n=68, 98) | 2.9 | 0.0

ADVERSE EVENTS:
Time Frame: Group 1: Baseline up to Day 280; Group 2, 3 and 4: Baseline up to Day 210. Participants recorded pre-specified AEs in electronic diary:local reactions; systemic events (up to 7 days after each vaccine dose)
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on the case report form at each visit (nonsystematic assessment).
Groups:
- 13vPnC Group 1 (Cohort 1) Dose 1; 13vPnC Group 2 (Cohort 1) Dose 1: 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to protocol amendment to increase sample size (Cohort 1).
- 13vPnC Group 1 (Cohort 1) Dose 2: 13vPnC (0.5mL dose) administered intramuscularly anytime from Day 56 to Day 70. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled prior to protocol amendment to increase sample size (Cohort 1).
- 13vPnC Group 1 (Cohort 2) Dose 1; 13vPnC Group 2 (Cohort 2) Dose 1: 13vPnC (0.5mL dose) administered intramuscularly at baseline. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled after protocol amendment to increase sample size (Cohort 2).
- 13vPnC Group 1 (Cohort 2) Dose 2: 13vPnC (0.5mL dose) administered intramuscularly anytime from Day 56 to Day 70. Participants must have previously received at least 3 doses of 7vPnC. Includes participants enrolled after protocol amendment to increase sample size (Cohort 2).
- 6-Month Follow-up 13vPnC Group 1 (Cohort 1 and 2): 6-month follow-up telephone contact for participants in Group 1 (Cohort 1 and 2).
- 6-Month Follow-up 13vPnC Group 2 (Cohort 1 and 2): 6-month follow-up telephone contact for participants in Group 2 (Cohort 1 and 2).
- 6-Month Follow-up 13vPnC Group 3: 6-month follow-up telephone contact for participants in Group 3.
- 6-Month Follow-up 13vPnC Group 4: 6 -Month Follow-up Telephone Contact for participants in Group 4.
Arm/Group | 13vPnC Group 1 (Cohort 1) Dose 1 | 13vPnC Group 1 (Cohort 1) Dose 2 | 13vPnC Group 2 (Cohort 1) Dose 1 | 13vPnC Group 1 (Cohort 2) Dose 1 | 13vPnC Group 1 (Cohort 2) Dose 2 | 13vPnC Group 2 (Cohort 2) Dose 1 | 6-Month Follow-up 13vPnC Group 1 (Cohort 1 and 2) | 6-Month Follow-up 13vPnC Group 2 (Cohort 1 and 2) | 13vPnC Group 3 | 6-Month Follow-up 13vPnC Group 3 | 13vPnC Group 4 | 6-Month Follow-up 13vPnC Group 4
Serious Adverse Events (participants affected / at risk) | 0/124 | 2/112 | 1/179 | 1/175 | 4/165 | 0/118 | 3/299 | 1/297 | 1/294 | 0/294 | 0/298 | 1/298
Other Adverse Events (participants affected / at risk) | 112/124 | 91/112 | 158/179 | 165/175 | 137/165 | 107/118 | 2/299 | 2/297 | 242/294 | 7/294 | 258/298 | 4/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Group 1 (Cohort 1) Dose 1 (N=124) | 13vPnC Group 1 (Cohort 1) Dose 2 (N=112) | 13vPnC Group 2 (Cohort 1) Dose 1 (N=179) | 13vPnC Group 1 (Cohort 2) Dose 1 (N=175) | 13vPnC Group 1 (Cohort 2) Dose 2 (N=165) | 13vPnC Group 2 (Cohort 2) Dose 1 (N=118) | 6-Month Follow-up 13vPnC Group 1 (Cohort 1 and 2) (N=299) | 6-Month Follow-up 13vPnC Group 2 (Cohort 1 and 2) (N=297) | 13vPnC Group 3 (N=294) | 6-Month Follow-up 13vPnC Group 3 (N=294) | 13vPnC Group 4 (N=298) | 6-Month Follow-up 13vPnC Group 4 (N=298)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Group 1 (Cohort 1) Dose 1 (N=124) | 13vPnC Group 1 (Cohort 1) Dose 2 (N=112) | 13vPnC Group 2 (Cohort 1) Dose 1 (N=179) | 13vPnC Group 1 (Cohort 2) Dose 1 (N=175) | 13vPnC Group 1 (Cohort 2) Dose 2 (N=165) | 13vPnC Group 2 (Cohort 2) Dose 1 (N=118) | 6-Month Follow-up 13vPnC Group 1 (Cohort 1 and 2) (N=299) | 6-Month Follow-up 13vPnC Group 2 (Cohort 1 and 2) (N=297) | 13vPnC Group 3 (N=294) | 6-Month Follow-up 13vPnC Group 3 (N=294) | 13vPnC Group 4 (N=298) | 6-Month Follow-up 13vPnC Group 4 (N=298)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 2 | 4 | 2 | 2 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 4 | 6 | 3 | 2 | 0 | 0 | 3 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 1 | 1 | 2 | 3 | 3 | 0 | 0 | 8 | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 3 | 3 | 7 | 5 | 4 | 0 | 0 | 7 | 0 | 3 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 15 | 5 | 12 | 12 | 11 | 1 | 0 | 0 | 3 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 9 | 3 | 15 | 14 | 1 | 0 | 0 | 2 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1 | 7 | 2 | 3 | 0 | 0 | 3 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 3 | 3 | 4 | 4 | 1 | 2 | 0 | 0 | 3 | 0 | 5 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 2 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 2 | 1 | 5 | 4 | 3 | 3 | 0 | 0 | 3 | 0 | 4 | 0
Croup infectious (Infections and infestations) | 2 | 1 | 2 | 7 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 5 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 5 | 0
Lice infestation (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Intertrigo candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 10 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asperger's disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 7 | 6 | 7 | 3 | 0 | 0 | 10 | 0 | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4 | 5 | 4 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 55/108 | 50/87 | 96/155 | 67/148 | 69/125 | 64/102 | 0/0 | 0/0 | 230/265 | 0/0 | 252/283 | 0/0
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 7/92 | 6/68 | 15/141 | 7/133 | 10/101 | 12/92 | 0/0 | 0/0 | 43/221 | 0/0 | 106/242 | 0/0
Swelling (any) (Skin and subcutaneous tissue disorders) | 25/97 | 17/73 | 32/144 | 25/142 | 18/105 | 18/90 | 0/0 | 0/0 | 85/226 | 0/0 | 86/233 | 0/0
Swelling (mild) (Skin and subcutaneous tissue disorders) | 20/94 | 16/72 | 29/143 | 20/141 | 16/104 | 12/89 | 0/0 | 0/0 | 48/220 | 0/0 | 50/221 | 0/0
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 9/94 | 2/69 | 8/141 | 10/135 | 8/102 | 10/89 | 0/0 | 0/0 | 48/219 | 0/0 | 48/226 | 0/0
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/90 | 0/68 | 0/138 | 0/131 | 0/98 | 1/88 | 0/0 | 0/0 | 7/211 | 0/0 | 4/214 | 0/0
Redness (any) (Skin and subcutaneous tissue disorders) | 41/103 | 27/76 | 52/149 | 27/143 | 26/110 | 33/91 | 0/0 | 0/0 | 100/233 | 0/0 | 70/232 | 0/0
Redness (mild) (Skin and subcutaneous tissue disorders) | 31/99 | 25/74 | 46/146 | 24/143 | 20/108 | 28/90 | 0/0 | 0/0 | 63/226 | 0/0 | 48/226 | 0/0
Redness (moderate) (Skin and subcutaneous tissue disorders) | 12/94 | 5/70 | 14/142 | 8/135 | 6/100 | 13/89 | 0/0 | 0/0 | 48/218 | 0/0 | 31/221 | 0/0
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/90 | 0/68 | 0/138 | 1/131 | 0/98 | 1/88 | 0/0 | 0/0 | 7/212 | 0/0 | 4/213 | 0/0
Fever >=38 degreesC but <=39 degreesC (General disorders) | 15/92 | 10/70 | 7/138 | 24/137 | 12/101 | 13/90 | 0/0 | 0/0 | 9/212 | 0/0 | 11/214 | 0/0
Fever >39 degreesC but <=40 degreesC (General disorders) | 4/90 | 3/68 | 1/138 | 6/130 | 2/100 | 3/89 | 0/0 | 0/0 | 5/212 | 0/0 | 1/212 | 0/0
Fever >40 degreesC (General disorders) | 0/90 | 0/68 | 1/138 | 0/130 | 1/98 | 1/88 | 0/0 | 0/0 | 1/210 | 0/0 | 1/212 | 0/0
Decreased appetite (General disorders) | 42/99 | 31/77 | 37/149 | 58/146 | 39/113 | 32/94 | 0/0 | 0/0 | 52/227 | 0/0 | 51/223 | 0/0
Irritability (General disorders) | 65/108 | 56/86 | 60/151 | 113/156 | 77/126 | 53/102 | 0/0 | 0/0 | 73/234 | 0/0 | 59/234 | 0/0
Increased sleep (General disorders) | 32/98 | 22/75 | 23/145 | 54/146 | 26/109 | 23/97 | 0/0 | 0/0 | 48/226 | 0/0 | 61/229 | 0/0
Decreased sleep (General disorders) | 22/97 | 22/77 | 20/143 | 45/140 | 30/112 | 17/91 | 0/0 | 0/0 | 12/212 | 0/0 | 42/224 | 0/0
Hives (urticaria) (General disorders) | 1/90 | 2/68 | 1/139 | 2/131 | 0/98 | 4/88 | 0/0 | 0/0 | 4/213 | 0/0 | 3/214 | 0/0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uvulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.